CLINICAL TRIAL: NCT06180330
Title: The Impact of Water Activities on Motor Development in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01-47/2023
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-12

CONDITIONS: Infant Development
Keywords: swimming; motor development; infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic baby class (Experimental): 8 weeks program of aquatic exercises for infants
  Interventions: Other: Aquatic baby class
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Other: Aquatic baby class — The intervention will consist of exercises for infants. They will be in the water together with parents
  Arms: Aquatic baby class

SUMMARY:
The study will be conducted at various city swimming pools in Warsaw. The study participants will include 20 infants participating in aquatic baby classes once a week and 20 infants not participating in any classes and their parents. The study will be conducted in a quiet and calm room, which will be prepared in advance and equipped with a smooth mat, a lounger and infant toys. The estimated time to conduct the study is about 30 minutes.

The examination will be carried out twice: before the start of the two-month course and after its completion. Each time in the presence of a parent or legal guardian, after signing a consent form for the study.

The selected methods of assessing motor development are fully non-invasive and consist of the following tests:

1. Alberta Infant Motor Scale (AIMS)-a test involving observation of motor development, in which each activity is assessed as existing or not. The sum of the scores from all trials is then placed on a centile grid, the results of which will indicate how many children of a certain age are achieving a given level of motor skills.
2. Early Motor Development Questionnaire (EMQ)-will be conducted on the basis of a ready-made form and in an anonymous manner based on parents' current knowledge of their children's development.

ELIGIBILITY:
Inclusion Criteria:

* infants age 3-12 months

Exclusion Criteria:

* any disability that would affect motor development

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Alberta Infant Motor Scale (AIMS) at 8 weeks | Baseline and 8 weeks
  The test involving observation of motor development, in which each activity is assessed as existing or not. The sum of the scores from all trials is then placed on a centile grid, the results of which will indicate how many children of a certain age are achieving a given level of motor skills.
  During the assessment, the evaluator observes the movements of the child and scores each movement component as either "observed" or "not observed".
Change from Baseline in the Early Motor Development Questionnaire (EMQ) at 8 weeks | Baseline and 8 weeks
  The questionnaire will be conducted on the basis of a ready-made form and in an anonymous manner based on parents' current knowledge of their children's development.
  EMQ incorporates parents' certainty in their answers by using a 5-point scale ranging from -2 (the parent is sure the child does not show the behavior yet) to +2 (the parent remembers a particular instance in which the child exhibited the behavior).

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw, Warsaw, Poland